CLINICAL TRIAL: NCT02341014
Title: Phase Ib/IIa Study of Combination Therapy With Carfilzomib, Romidepsin, Lenalidomide in Patients With Relapsed or Refractory B- and T-cell Lymphomas
Brief Title: Combination Therapy With Carfilzomib, Romidepsin, Lenalidomide in Patients With Relapsed or Refractory B- and T-cell Lymphomas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-179
Record Dates: First submitted 2015-01-14; First posted 2015-01-19 (Estimated); Results first posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2023-01

CONDITIONS: T-cell Lymphomas; Relapsed or Refractory
Keywords: Carfilzomib; Romidepsin; Lenalidomide; Lymphomas; 14-179
MeSH Terms: conditions — Lymphoma, T-Cell; Recurrence; Lymphoma | interventions — carfilzomib; romidepsin; Lenalidomide

ARMS (1):
- Carfilzomib, Romidepsin, Lenalidomide (Experimental): All patients will be treated with romidepsin administered intravenously on days 1 and 8 of a 21-day cycle. Lenalidomide will be taken orally daily for days 1-14 of a 21-day cycle. The carfilzomib will be given weekly on days 1, and 8 of a 21-day cycle.
  Interventions: Drug: Carfilzomib; Drug: Romidepsin; Drug: Lenalidomide

INTERVENTIONS:
Drug: Carfilzomib — The initial dose of carfilzomib (cycle 1, day 1) given to any patient must be 20mg/m2 .
Drug: Romidepsin
Drug: Lenalidomide

SUMMARY:
This is an open label phase Ib/IIa study of patients with relapsed/refractory B- and T-cell lymphomas who are treated with carfilzomib, lenalidomide and romidepsin.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed B- or T-cell lymphomas at the enrolling institution, including stage ≥ Ib CTCL, which has relapsed or progressed after at least one systemic therapy.
* Hodgkin lymphoma is allowed and will be classified as a B-cell lymphoma in the phase IIA portion.
* Age ≥ 18,
* Previous systemic anti-cancer therapy must have been discontinued at least 3 weeks prior to treatment and adverse effects must have resolved to ≤Grade 1 or baseline. In the phase IIa portion, in progressing subjects, a 2 week washout may be allowed after discussion with the MSK Principal Investigator.
* Previous radiation, hormonal therapy, and/or surgery must have been discontinued or completed at least 2 weeks prior to treatment in this study and adverse effects must have resolved. Lymph node or other diagnostic biopsies within 2 weeks are not considered exclusionary.
* ECOG ≤ 2
* Meet the following laboratory criteria:
* Absolute neutrophil count 1.0/mm³,
* Platelet count 80 K/μ (in the Phase II portion, if thrombocytopenia is due to bone marrow involvement platelet count must be 50 K/μL),
* Phase Ib subjects must have calculated creatinine clearance 50ml/min by Cockcroft-Gault formula, phase IIa subjects must have calculated creatinine clearance ≥ 40ml4/min by Cockcroft-Gault formula.
* Total bilirubin 1.5 x upper limit of normal (ULN); AST (SGOT) and ALT (SGPT) 3 x ULN
* Measurable disease for phase IIa portion only.
* Lymphoma (includes CTCL patients who are without evidence of the disease in the skin): CT or PET/CT by modified Cheson criteria with incorporation of PET.
* CTCL: mSWAT >0, or absolute Sezary count ≥ 1000 cells/μL.
* All study participants must be registered into the mandatory Revlimid REMS ® program, and be willing and able to comply with the requirements of the REMS ® program.
* Short course systemic corticosteroids for disease control, improvement of performance status or non-cancer indication (< 7 days) must have been discontinued at least 6 days prior to study treatment. Stable ongoing corticosteroid use (≥ 30 days) up to an equivalent dose of 15 mg of prednisone is permissible.
* Topical steroids that have been used for > 3 weeks may be continued (CTCL only).
* Women of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS® program. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. See Appendix A: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods.
* A female of reproductive potential is a sexually mature female who:
* has not undergone a hysterectomy or bilateral oophorectomy; or has not been naturally postmenopausal for at least 24 consecutive months (i.e. has had menses at any time in the preceding 24 consecutive months).

Exclusion Criteria:

* Patients who have a standard curative option for their lymphoid malignancy at current state of disease are excluded. For eligibility on this trial, allogeneic stem cell transplantation is not to be considered a standard curative option.
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant females. (Lactating females must agree not to breast feed while taking carfilzomib, lenalidomide or romidepsin).
* Known hypersensitivity to thalidomide.
* The development of erythema multiforme if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Prior use of lenalidomide if discontinued due to toxicity.
* Prior therapy with romidepsin if discontinued due to toxicity.
* Prior therapy with carfilzomib if discontinued due to toxicity.
* Prior therapy with a proteasome inhibitor if discontinued due to toxicity.
* Concurrent use of other anti-cancer agents or treatments.
* Known seropositive and requiring anti-viral therapy for human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV).
* Concurrent malignancy requiring active therapy.
* Patients with more than one type of lymphoma may be enrolled after discussion with the MSK Principal Investigator.
* Known central nervous system or meningeal involvement (in the absence of symptoms investigation into central nervous system involvement is not required).
* The following known cardiac abnormalities:
* Congenital long QT syndrome.
* QTc/QTf interval ≥ 480 milliseconds; unless secondary to pacemaker or bundle branch block.
* Myocardial infarction within 6 months of cycle one, day one (C1D1). Subjects with a history of myocardial infarction between 6 and 12 months prior to C1D1 who are asymptomatic and have had a negative cardiac risk assessment (treadmill stress test, nuclear medicine stress test, or stress echocardiogram) since the event may participate.
* Other significant ECG abnormalities including 2nd degree atrio-ventricular (AV) block type II, 3rd degree AV block.
* Symptomatic coronary artery disease (CAD), e.g., angina Canadian Class II-IV (see Appendix B). In any patient in whom there is doubt, the patient should have a stress imaging study and, if abnormal, angiography to define whether or not CAD is present.
* An ECG recorded at screening showing evidence of cardiac ischemia (ST depression of ≥2 mm, measured from isoelectric line to the ST segment). If in any doubt, the patient should have a stress imaging study and, if abnormal, angiography to define whether or not CAD is present.
* Congestive heart failure (CHF) that meets New York Heart Association (NYHA) Class II to IV definitions (see Appendix C) and/or ejection fraction <45% by, echocardiogram, or cardiac MRI.
* A known history of sustained ventricular tachycardia (VT), ventricular fibrillation (VF), Torsade de Pointes, or cardiac arrest unless currently addressed with an automatic implantable cardioverter defibrillator (AICD).
* Hypertrophic cardiomegaly or restrictive cardiomyopathy from prior treatment or other causes.
* Uncontrolled hypertension, i.e., blood pressure (BP) of ≥170/95; patients who have a history of hypertension controlled by medication must be on a stable dose (for at least one month) and meet all other inclusion criteria.
* Any cardiac arrhythmia requiring an anti-arrhythmic medication (excluding stable doses of beta-blockers)
* Patients taking drugs that can cause significant QTc/QTf prolongation unless able to be switched to non-QTc/QTf prolonging medication or on a stable dose without significant QT prolongation (>470 msec).
* Concomitant use of significant CYP3A4 inhibitors unless able to be switched to a non-CYP3A4 inhibiting medication.
* Caution should be used when administering study drugs to patients taking medications significantly metabolized by these enzymes refer to (http://medicine.iupui.edu/clinpharm/ddis/clinical-table/ ) for clinically relevant medications. Particular attention should be paid to patients receiving warfarin. Patient should have coagulation parameters monitored regularly, and warfarin dose adjusted accordingly. If these drugs cannot be discontinued or replaced, enrollment may be allowed after discussion with MSK PI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-01-02 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Horwitz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase Ib: DL 1; Phase IIa - MTD: Romidepsin (8mg/m2 IV) + Lenalidomide (15mg PO, QD) + Carfilzomib (36 mg/m2 IV)
- Phase Ib: DL 2: Romidepsin (8mg/m2 IV) + Lenalidomide (15mg PO, QD) + Carfilzomib (45 mg/m2 IV)
- Phase Ib: DL 3: Romidepsin (10mg/m2 IV) + Lenalidomide (20mg PO, QD) + Carfilzomib (45 mg/m2 IV)
- Phase Ib: DL 4: Romidepsin (10mg/m2 IV) + Lenalidomide (20mg PO, QD) + Carfilzomib (56 mg/m2 IV)
Period: Overall Study
Arm/Group | Phase Ib: DL 1 | Phase Ib: DL 2 | Phase Ib: DL 3 | Phase Ib: DL 4 | Phase IIa - MTD
Started | 6 | 7 | 0 | 0 | 14
Completed | 6 | 6 | 0 | 0 | 12
Not Completed | 0 | 1 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: MTD was established after Dose Level/DL 2 so no participants were treated on DL 3 or DL 4
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase Ib: DL 1 | Phase Ib: DL 2 | Phase Ib: DL 3 | Phase Ib: DL 4 | Phase IIa - MTD | Total
Number analyzed (Participants) | 6 | 7 | 0 | 0 | 14 | 27
Age, Continuous [Median (Full Range); unit: years] | 60 [44 to 66] | 67 [44 to 74] |  |  | 56 [36 to 83] | 57 [36 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 |  |  | 2 | 6
  Male | 4 | 5 |  |  | 12 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 |  |  | 0 | 1
  Not Hispanic or Latino | 5 | 7 |  |  | 11 | 23
  Unknown or Not Reported | 0 | 0 |  |  | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  |  | 0 | 0
  Asian | 1 | 0 |  |  | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  | 0 | 0
  Black or African American | 1 | 0 |  |  | 0 | 1
  White | 4 | 7 |  |  | 13 | 24
  More than one race | 0 | 0 |  |  | 0 | 0
  Unknown or Not Reported | 0 | 0 |  |  | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 7 |  |  | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Romidepsin
Description: Determine the MTD by NCI-CTCAE v4.0.
Time Frame: 21 days
Population: Phase Ib participants
Measure: Number; unit: mg/m^2 romidepsin
Arm/Group | Phase Ib: DL 1 | Phase Ib: DL 2
Number analyzed (Participants) | 6 | 7
mg/m^2 romidepsin | 8 | 8

2. Primary Outcome: Maximum Tolerated Dose of Lenalidomide
Description: Determine the MTD by NCI-CTCAE v4.0.
Time Frame: 21 days
Population: Phase Ib participants
Measure: Number; unit: mg of Lenalidomide
Arm/Group | Phase Ib: DL 1 | Phase Ib: DL 2
Number analyzed (Participants) | 6 | 7
mg of Lenalidomide | 15 | 15

3. Primary Outcome: Maximum Tolerated Dose of Carfilzomib
Description: Determine the MTD by NCI-CTCAE v4.0.
Time Frame: 21 days
Population: Phase Ib participants
Measure: Number; unit: mg/m^2 of Carfilzomib
Groups:
- Phase 1b: DL 1: Romidepsin (8mg/m2 IV) + Lenalidomide (15mg PO, QD) + Carfilzomib (36 mg/m2 IV)
- Phase 1b: DL 2: Romidepsin (8mg/m2 IV) + Lenalidomide (15mg PO, QD) + Carfilzomib (45 mg/m2 IV)
Arm/Group | Phase 1b: DL 1 | Phase 1b: DL 2
Number analyzed (Participants) | 6 | 7
mg/m^2 of Carfilzomib | 36 | 36

4. Secondary Outcome: Overall Response Rate (Orr) at the Maximum Tolerated Dose
Description: will be summarized using percentages and confidence intervals will be provided. ORR will be calculated based on the best response at any time during the course of treatment on this protocol.
Time Frame: 1 year
Population: T-cell Lymphoma participants evaluable for response at the maximum tolerated dose
Measure: Number (95% Confidence Interval); unit: percentage of pts with response
Arm/Group | Phase 1b: DL 1 | Phase 1b: DL 2 | Phase IIa - MTD
Number analyzed (Participants) | 6 | 7 | 14
percentage of pts with response | 50 [12 to 88] | 57 [18 to 90] | 42 [15 to 72]

ADVERSE EVENTS:
Time Frame: 1 year
Description: Participants were not enrolled on Dose Level/DL 3 and DL4.
Arm/Group | Phase Ib: DL 1 | Phase Ib: DL 2 | Phase Ib: DL 3 | Phase Ib: DL 4 | Phase IIa - MTD
All-Cause Mortality (participants affected / at risk) | 4/6 | 6/7 | 0/0 | 0/0 | 8/14
Serious Adverse Events (participants affected / at risk) | 0/6 | 5/7 | 0/0 | 0/0 | 3/14
Other Adverse Events (participants affected / at risk) | 2/6 | 6/7 | 0/0 | 0/0 | 5/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase Ib: DL 1 (N=6) | Phase Ib: DL 2 (N=7) | Phase Ib: DL 3 (N=0) | Phase Ib: DL 4 (N=0) | Phase IIa - MTD (N=14)
Anemia (Blood and lymphatic system disorders) | 0 | 1 | NA | NA | 0
Chills (General disorders) | 0 | 0 | NA | NA | 1
Death NOS (General disorders) | 0 | 0 | NA | NA | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | NA | NA | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | NA | NA | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | NA | NA | 1
Edema (General disorders) | 0 | 1 | NA | NA | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | NA | NA | 1
Fever (General disorders) | 0 | 2 | NA | NA | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA | 0
Heart failure (Cardiac disorders) | 0 | 0 | NA | NA | 1
Hypotension (Vascular disorders) | 0 | 0 | NA | NA | 1
Lung infection (Infections and infestations) | 0 | 0 | NA | NA | 1
Thromboembolic event (Vascular disorders) | 0 | 1 | NA | NA | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | NA | NA | 0
Thrombocytopenia (Investigations) | 0 | 1 | NA | NA | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase Ib: DL 1 (N=6) | Phase Ib: DL 2 (N=7) | Phase Ib: DL 3 (N=0) | Phase Ib: DL 4 (N=0) | Phase IIa - MTD (N=14)
Anemia (Blood and lymphatic system disorders) | 0 | 2 | NA | NA | 0
Platelet count decreased (Investigations) | 1 | 3 | NA | NA | 2
White blood cell decreased (Investigations) | 0 | 2 | NA | NA | 1
Neutrophil count decreased (Investigations) | 1 | 4 | NA | NA | 2
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | NA | NA | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | NA | NA | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0 | NA | NA | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | NA | NA | 1
Weight loss (Investigations) | 0 | 2 | NA | NA | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-06): https://cdn.clinicaltrials.gov/large-docs/14/NCT02341014/Prot_SAP_000.pdf